CLINICAL TRIAL: NCT05497102
Title: Phase II, Single-arm Trial of Carfilzomib, Lenalidomide, and Dexamethasone Re-induction Followed by the 2nd ASCT in Multiple Myeloma Patients Relapsed After the 1st ASCT
Brief Title: Carfilzomib, Lenalidomide, and Dexamethasone Re-induction Followed by the 2nd ASCT in Multiple Myeloma Patients Relapsed After the 1st ASCT
Acronym: KMM1911
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Kihyun Kim, Professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMC 2019-12-037
Record Dates: First submitted 2022-07-27; First posted 2022-08-11 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm of Lenalidomide maintenance (Experimental): [KRd #1~6, Every 4 weeks] D1, 2, 8, 9, 15,16 Carfilzomib 20mg/m2 + 5% dextrose in water 50 mL over 10 mins (From Cycle1Day8 27mg/m2) D1 - 21 Lenalidomide 25mg P.O. D1, 8, 15, 22 Dexamethasone 40mg IV or PO
  [Autologous stem cell transplantation phase]
  [Lenalidomide maintenance phase, Every 4 weeks] D1-28 Lenalidomide 10 mg
  Interventions: Drug: Lenalidomide maintenance

INTERVENTIONS:
Drug: Lenalidomide maintenance — Lenalidomide maintenance after carfilzomib, lenalidomide, and dexamethasone re-induction followed by the 2nd ASCT.

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of salvage treatment with carfilzomib/lenalidomide/dexamethasone (KRD) followed by 2nd autologous stem cell transplantation (ASCT) and lenalidomide maintenance in patients with relapsed myeloma after 1st ASCT.

DETAILED DESCRIPTION:
This is a single-arm phase II study to assess the efficacy and safety of KRD followed by 2nd ASCT - lenalidomide maintenance for 18 months in patients with relapsed multiple myeloma after 1st ASCT who are 70 years of age or younger. A total of 58 participants will be recruited. As a re-induction therapy 6 cycles of KRD (K, 27mg/m2, D1,2,8,9,15,16; R, 25 mg, D1-21; D, 40mg weekly, every 28 days) will be administered. If a patient achieves at least partial response, 2nd ASCT + lenalidomide 10mg for 18 months will be proceeded. Study will be continued until disease progression, unacceptable toxicity, or completion of pre-planned schedule. Response will be assessed using the International Myeloma Working Group(IMWG) response criteria and the safety profiles will be described using the NCI-CTCAE v5.0. Participants who discontinue therapy will be followed every 3 months for 3 years if they are on subsequent treatment, disease-free or dead.

ELIGIBILITY:
Inclusion Criteria:

1. Age 20~70
2. Progressive disease after 1st ASCT
3. Duration of response after 1st ASCT > 12 months
4. Measurable disease (+)

   * Serum M-protein ≥ 1 g/dL
   * Urine M-protein ≥ 200 mg/24 hr
   * Serum Free Light Chain(FLC) assay: involved FLC level ≥10 mg/dL (serum Free Light Chain ratio is abnormal)
5. Adequate organ function for induction & ASCT

   * Absolute Neutrophil Count (ANC) ≥ 1.0 x 109/L
   * Platelets ≥ 50 x 109/L (≥ 30 x 109/L if myeloma involvement is > 50% in the bone marrow)
   * Hemoglobin ≥ 8.0 g/dL
   * Creatinine clearance ≥ 30 mL/minute
   * Serum Bilirubin ≤ 1.5 x upper limit of normal
   * Aspartate aminotransferase(AST) and Alanine aminotransferase(ALT) ≤ 3 x upper limit of normal
6. Eastern Cooperative Oncology Group performance scale 0~2
7. Survival expectancy > 3 months
8. Adequately controlled hepatitis B(HBV) & hepatitis C(HCV)
9. Written informed consent
10. Optimal contraceptions

Exclusion Criteria:

1. Prior refractoriness or intolerance to carfilzomib
2. Prior refractoriness or intolerance to lenalidomide/dexamethasone
3. Any treatment after progressive disease after 1st ASCT. High-dose dexamethasone or palliative radiation is permitted.
4. Waldenstroem's macroglobulinemia, POEMS syndrome, or plasma cell leukemia
5. Pregnant or nursing lactating women
6. Myocardial infarct within 6 months, heart failure of New York Heart Association(NYHA) Class III~IV, uncontrolled ventricular arrhythmia, severe coronary arterial obstructive disease
7. Uncontrolled hypertension (Defined as an average systolic blood pressure >= 160 mmHg or diastolic >= 100 mmHg) or diabetes
8. Grade 3~4 neuropathy
9. HIV infection
10. Severe or uncontrolled medical conditions, laboratory abnormalities, or psychiatric disorders that may preclude the participation of the study by the physician's discretion
11. Contraindication to any of the required concomitant drugs or supportive treatments, including hypersensitivity to all anticoagulation and antiplatelet options, antiviral drugs, or intolerance to hydration due to preexisting pulmonary or cardiac impairment
12. Diagnosis of other malignant disease other than myeloma within 5 year. Exceptions are properly treated non-melanomatous skin cancers, cervical intraepithelial neoplasia, prostate cancer that do not require treatment, or properly excised well-differentiated thyroid cancers

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2021-11-08 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
2-year progression free survival rate | 2-years after the written consent
  percentage of patients who are disease free or alive at 2-years

SECONDARY OUTCOMES:
Complete response rate after KRd #6 | total 6 cycles (each cycle is 28 days) of induction therapy
  percentage of patients who achieve complete response
Complete response rate after ASCT | at the time of 2nd ASCT (within 60 days after ASCT)
  percentage of patients who achieve complete response
Overall response rate | assessed for approximately 3 years after administration
  percentage of patients who achieve at least partial response
Time to response | assessed for approximately 3 years after administration
  from the time of written consent to the time of achieving at least partial response
Duration of response | assessed for approximately 3 years after administration
  from the time of achieving at least partial response to the time of progressive disease
Overall survival | assessed for approximately 3 years after administration
  from the time of written consent to the time of death or last follow-up
Safety of KRd induction therapy, 2nd ASCT, and lenalidomide maintenance therapy | assessed for approximately 2 years during administration
  treatment-emergent adverse events
Rate of the successful stem cell harvest | total 6 cycles (each cycle is 28 days) of induction therapy
  percentage of patients who collected cluster of differentiation(CD34+) hematopoietic stem cells > 2 x 10^6 cells/kg

CONTACTS AND LOCATIONS:
Overall Officials: Kihyun Kim, M.D., Ph.D, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided